CLINICAL TRIAL: NCT03408795
Title: Assessing the Surgical Skills of Trainees in Learning the Laparoscopic Distal Gastrectomy
Brief Title: Assessing the Surgical Skills of Trainees in Learning the LDG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nagasaki University (Other)
Collaborators: Hokkaido University (Other)
Responsible Party: Principal Investigator, Kobayashi Shinichiro, Principal Investigator, Department of Surgery, Nagasaki University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15122118
Record Dates: First submitted 2018-01-08; First posted 2018-01-24 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Gastrostomy; Surgical Procedure, Unspecified; Assessment, Self

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JORS-LDG Group (Other): Participants in JORS-LDG Group score the performance of procedure after LDG.
  Interventions: Procedure: Laparoscopic distal gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic distal gastrectomy — Longitudinal testing of The Japanese Operative Rating Scale for Laparoscopic Distal Gastrectomy

SUMMARY:
Laparoscopic distal gastrectomy (LDG) is a common surgery in the surgical trainees. However, there is no assessment system to measuring the surgical skill of surgical trainees. The novel surgical assessment system, which called Japanese Operative Rating Scale for Laparoscopic Distal Gastrectomy (JORS-LDG) by the task analysis and the Delphi method have been developed. This study describes assessing the development of surgical skill by JORS-LDG in the initial experience of LDG.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic distal gastrectomy to early gastric cancer
* D1 plus or D2 lymphadenectomy
* Provide signed informed consent

Exclusion Criteria:

* postoperative conditions affecting LDG
* pregnancy
* advanced gastric cancer
* D1 lymphadenectomy
* Total or subtotal gastrectomy
* unsuitable condition

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Assessing the development of surgical skill by JORS-DG in the initial experience of LDG. | Participants will be followed for the duration of the educational study for 3 years.
  The surgical skill and performance of LDG was scored using JORS-DG by a trainee and an instructor. The difference in mean surgical performance score of JORS-DG was evaluated in tree phase. The score about JORS-DG is evaluated on a three or two level scale ( 28items in B-1 reconstruction or 31items in R-Y reconstruction). Maximum of total score is 46 in B-1 reconstruction or 52 in R-Y reconstruction. High score is good surgical skill. Low score is poor surgical skill.

SECONDARY OUTCOMES:
Assessing the value of surgical skill by JORS-DG in the initial experience of LDG and surgical outcome. | Participants will be followed for the duration of the educational study for 3 years.
  Operation time, bleeding , Postoperative complications are compared with average of total score of JORS-LDG. The score about JORS-LDG is evaluated on a three or two level scale ( 28items in B-1 reconstruction or 31items in R-Y reconstruction). Maximum of total score is 46 in B-1 reconstruction or 52 in R-Y reconstruction. High score is good surgical skill. Low score is poor surgical skill.
Assessing the value of surgical skill by JORS-DG in the initial experience of LDG and surgical outcome. | Participants will be followed for the duration of the educational study for 3 years.
  Procedures' time in each items of LDG was evaluated for difficulty of surgical technics. The scoring rates in each items of LDG are compared with Procedures' time. The average of score about JORS-LDG is evaluated on a three or two level scale ( 28items in B-1 reconstruction or 31items in R-Y reconstruction). High score is good surgical skill. Low score is poor surgical skill.

CONTACTS AND LOCATIONS:
Locations (1):
- Nagasaki University Hospital, Nagasaki, Japan

IPD SHARING:
Plan to Share IPD: No